CLINICAL TRIAL: NCT06358846
Title: Effectiveness of Educational Intervention on Footcare Among Individuals Having Type 2 Diabetes at Slums of Karachi, Pakistan. A Randomize Control Trial.
Brief Title: Effectiveness of Educational Intervention on Footcare Among Individuals Having Type 2 Diabetes at Slums of Karachi, Pakistan.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: SINA Health Education and Welfare Trust (Other)
Collaborators: Aga Khan University (Other)
Responsible Party: Principal Investigator, Hina Sharif, Assistant Manager, SINA Health Education and Welfare Trust
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 00004
Record Dates: First submitted 2024-04-07; First posted 2024-04-11 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Diabetic Foot; Educational Intervention; Foot Care; Foot Ulcer, Diabetic; Foot Cellulitis
Keywords: Type 2 Diabetes; slums population; vulnerable population; low-socioeconomic status; Diabetes foot care; Knowledge on foot care
MeSH Terms: conditions — Diabetic Foot; Diabetes Mellitus, Type 2

STUDY DESIGN:
Intervention Model Description: Control arm =75 Interventional arm = 75
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- standard care advice (No Intervention): The control group will simply get standard advice from clinicians at the clinic during consultations.
- standard care advice+ structured training through pictures containing learning pamphlet (Experimental): Interventional group will receive standard advice from clinician along with the structured training from qualified diabetes' educator through pictures containing learning pamphlet
  Interventions: Behavioral: Self-care behavior to promote foot care through educational guidance among individual with diabetes

INTERVENTIONS:
Behavioral: Self-care behavior to promote foot care through educational guidance among individual with diabetes — Apart from physician consultation, individuals will received structured training of how to care their foot to avoid ulcer and inflammation.
  Arms: standard care advice+ structured training through pictures containing learning pamphlet

SUMMARY:
There are multiple studies conducted in Pakistan that supports the topic of foot care knowledge among individual with type 2 diabetes but all are descriptive cross-sectional studies and investigators cannot develop cause effect relationship out of it. Secondly, there is a lack of documented research on the foot care knowledge shown by people with T2D residing in the slums of Karachi. In order to assess the knowledge intervention among the individual having T2D through qualified diabetes educators and pictorial educational pamphlet along with the standard care of treatment. Consequently, it may aid in the development of effective methods aimed at mitigating foot-related complications among this specific population. Individuals diagnosed with diabetes are required to engage in proactive and structured self-care activities by providing the foot care knowledge in order to effectively manage their condition and mitigate the risk of potential complications. The incorporation of health-deviation knowledge and activities into routine is crucial.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients aged 18 years or older.
* Patients who are registered at designated SINA clinic and clinical and biochemical diagnosis of DM for at least six months
* Patients who are able to understand Urdu language will be included in the study
* Patients who are voluntarily participated the study will be included.

Exclusion Criteria:

* Patients come with recurrent foot ulcers or gangrene.
* History of amputation
* Patient live in other than designated slums location.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-08-15 (Actual); Study Completion 2024-08-31 (Actual)

PRIMARY OUTCOMES:
Improved Foot Care Knowledge | Time Frame: Three months after patient counselling towards foot care
  One potential outcome will be an increase in knowledge among participants regarding foot care practices specific to managing diabetes. This will include understanding the importance of proper footwear, regular foot inspections, and hygiene practices.
Behavior Change | Time Frame: Three months after patient counselling towards foot care
  The educational intervention will lead to positive changes in behavior related to foot care. Participants will be more likely to engage in recommended foot care practices such as daily foot inspections, avoiding walking barefoot, and seeking prompt medical attention for any foot-related issues.

SECONDARY OUTCOMES:
Reduction in Foot Complications | 3 months
  A successful educational intervention will potentially lead to a decrease in foot complications among individuals with Type 2 Diabetes. This will include a reduction in foot ulcers, infections, and amputations, ultimately improving participants' overall quality of life.
Empowerment and Self-efficacy | Three months treatment
  Participation in the educational intervention will empower individuals to take greater control of their diabetes management, leading to increased self-efficacy in managing their condition. This will result in improved confidence in their ability to prevent and manage foot complications.

CONTACTS AND LOCATIONS:
Locations (1):
- SINA Mewasha & North Clinic, Karachi, Sindh, Pakistan

REFERENCES:
- [Derived] Sharif H, Kadir M, Hashmi M, Naz S, Azam I, Imam A, Masood MQ. Effectiveness of pictorial educational intervention on foot care among individuals having type 2 diabetes at slums of Karachi, Pakistan: asingle blinded randomized control trial. BMC Public Health. 2025 Sep 30;25(1):3214. doi: 10.1186/s12889-025-23969-6. PMID 41029643